CLINICAL TRIAL: NCT05468606
Title: Coadministration of Genetically Attenuated Plasmodium Falciparum ∆mei2 (GA2) Sporozoites With Adjuvants - a Proof of Principle Study
Brief Title: Coadministration of GA2 Sporozoites With Adjuvants
Acronym: CoGA
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Meta Roestenberg, Prof. dr., Leiden University Medical Center
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: CoGA
Record Dates: First submitted 2022-07-14; First posted 2022-07-21 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Malaria,Falciparum
MeSH Terms: conditions — Malaria, Falciparum | interventions — Imiquimod

STUDY DESIGN:
Intervention Model Description: The study will consist of three stages (A, B, C). In stage A of the study, ten GA2 immunized participants will be compared to five infectivity controls in a blinded design. If the protective efficacy of the GA2 immunized group is ≤7/10 and some efficacy is seen in stage A (either ≥10% protection or significant increase in time to parasitemia) then the study will progress to stage B. In this stage, BCG (n=5), YF-17D (n=5) or imiquimod (n=5) will be applied/administered to the GA2 administration site. Additionally, two infectivity controls will participate in stage B.
  Based on the data on safety, tolerability and immunogenicity, the most favorable adjuvant of stage B can be chosen to be further assessed in stage C. In stage C, additional participants will be immunized with 50 GA2 infected mosquitoes in combination with the selected adjuvant. Additionally, a group of five unadjuvanted GA2 immunized participants and three infectivity controls will participate.
Who Masked: Participant, Investigator
Masking Description: Stage A will be randomized and double blind. Stage B will be open-label. The adjuvanted group of stage C will be open-label, the unadjuvanted group and the infectivity controls will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- GA2 group (unadjuvanted group) (Experimental): Immunization with 50 GA2-infected mosquito bites
  Interventions: Biological: GA2
- Infectivity controls (placebo group) (Placebo Comparator): Mock-immunization with 50 uninfected-mosquito bites
  Interventions: Other: Mock immunization
- BCG group (Experimental): Immunization with 50 GA2-infected mosquito bites and a standard intradermal BCG vaccination (0.1 mL)
  Interventions: Biological: GA2; Biological: BCG
- YF-17D group (Experimental): Immunization with 50 GA2-infected mosquito bites and a one fifth fractional (0.1 mL) intradermal YF-17D vaccination
  Interventions: Biological: GA2; Biological: YF-17D (fractional ID dose)
- Imiquimod group (Experimental): Immunization with 50 GA2-infected mosquito bites and 250mg imiquimod cream 5%
  Interventions: Biological: GA2; Drug: Imiquimod

INTERVENTIONS:
Biological: GA2 — GA2 sporozoites administered by 50 mosquito bites
  Arms: BCG group; GA2 group (unadjuvanted group); Imiquimod group; YF-17D group
Biological: BCG — 0.1 mL BCG vaccine intradermally
  Arms: BCG group
Biological: YF-17D (fractional ID dose) — 0.1 mL YF17D vaccine intradermally
  Other Names: Stamaril
  Arms: YF-17D group
Drug: Imiquimod — 250mg imiquimod 5% cream topical
  Other Names: Aldara
  Arms: Imiquimod group
Other: Mock immunization — 50 bites by uninfected mosquitoes
  Arms: Infectivity controls (placebo group)

SUMMARY:
This study will assess the coadministration of genetically attenuated Plasmodium falciparum ∆mei2 (GA2) sporozoites with adjuvants (BCG and YF-17D vaccination and imiquimod cream). Primary outcomes will be safety, tolerability and protective efficacy against CHMI.

DETAILED DESCRIPTION:
This will be an adaptive design single center, randomized controlled partly blinded, partly open-label clinical proof-of-principle trial of the genetically attenuated parasite GA2 co-administered with adjuvants in healthy, malaria-naïve male and female participants with no prior history of BCG or YF-17D vaccination. A total of 45 participants will be immunized by the bites of 50 GA2 infected mosquitos. Additionally, ten participants will serve as infectivity controls and will be exposed to the bites of 50 uninfected mosquitoes in the immunization phase.

During the 42 days following the immunization, there will be four out-patient visits and one phone call visit to evaluate adverse events and for hematology, biochemistry and immunology laboratory assessment. Six weeks after immunization, all 45 participants will undergo a CHMI through the bites of 5 mosquitos infected with wild-type 3D7 sporozoites. From day 6 to 21 after CHMI, participants will be followed daily on an out-patient basis to determine parasite loads detected by a quantitative polymerase chain reaction (qPCR). As soon as parasitemia is detected (cut-off >100p/mL), or at the latest 28 days after CHMI, participants will be treated with a curative regimen of antimalarials. The trial will be held in two cohorts: the second cohort starting 4 weeks after the first. The first cohort will consist of 10 participants and the second cohort will consist of 15 participants. Both cohorts will be block randomized to the five different study groups.

The study will consist of three stages. In stage A of the study, ten GA2 immunized participants will be compared to five infectivity controls in a blinded design. If the protective efficacy of the GA2 immunized group is ≤7/10 and some efficacy is seen in stage A (either ≥10% protection or significant increase in time to parasitemia) then the study will progress to stage B. In this stage, BCG (n=5), YF-17D (n=5) or imiquimod (n=5) will be applied/administered to the GA2 administration site. Additionally, two infectivity controls will participate in stage B. Stage B will be open label.

Based on the data on safety, tolerability and immunogenicity, the most favorable adjuvant of stage B can be chosen to be further assessed in stage C. In stage C, additional participants will be immunized with 50 GA2 infected mosquitoes in combination with the selected adjuvant. Additionally, a group of five unadjuvanted GA2 immunized participants and three infectivity controls will participate. The adjuvanted group of stage C will be open-label, the unadjuvanted group and the infectivity controls will be blinded.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is aged ≥18 and ≤35 years and in good health.
2. Participant has adequate understanding of the procedures of the study and agrees to abide strictly thereby.
3. Participant is able to communicate well with the investigator
4. Participant is available to attend all essential study visits.
5. Participant agrees that his/her general practitioner (GP) will be informed about participation in the study.
6. Participant agrees to refrain from blood donation to the national blood bank or for other purposes throughout the study period and for a defined period thereafter according to national blood bank guidelines.
7. Participants of child bearing potential (i.e., have an uterus and are neither surgically sterilized nor post-menopausal) agree to use adequate contraception and to not breastfeed for the duration of study.
8. Participant agrees to refrain from intensive physical exercise (disproportionate to the participants' usual daily activity or exercise routine) for twenty-one days following the immunization and during the malaria challenge period.
9. Participant signs informed consent.

   Exclusion Criteria:

   - 1. Any history, or evidence at screening, of clinically significant symptoms, physical signs or abnormal laboratory values suggestive of systemic conditions which could compromise the health of the participant during the study or interfere with the interpretation of the study results. These include, but are not limited to, any of the following:

   a. Body Mass Index (BMI) >35.0 kg/m2 at screening. b. An elevated risk of cardiovascular disease, defined as: i. An estimated ten-year risk of fatal cardiovascular disease of ≥5% at screening, as determined by the Systematic Coronary Risk Evaluation 2 (SCORE2) .

   ii. History, or evidence at screening, of clinically significant arrhythmia's, prolonged QT-interval or other clinically relevant ECG abnormalities; or iii. A positive family history of cardiac events in first- or second-degree relatives (according to the system used in medical genetics) <50 years old.

   c. Known functional asplenia, sickle cell trait/disease, thalassemia trait/disease or G6PD deficiency.

   d. History of epilepsy in the period of five years prior to study onset, even if no longer on medication.

   e. Positive HIV, HBV or HCV screening tests. f. Chronic use of i) immunosuppressive drugs, ii) antibiotics, iii) or other drugs that might have an influence on the immune system (excluding inhaled and topical corticosteroids and incidental use of oral anti-histamines), within three months prior to study onset or expected use of such during the study period.

   g. Skin disease affecting the site of administration in such a way that administration of mosquito bites or adjuvants is deemed impossible by investigator.

   h. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past five years.

   i. Any history of treatment for severe psychiatric disease by a psychiatrist in the past year.

   j. History of drug or alcohol abuse interfering with normal social functioning in the period of one year prior to study onset, positive urine toxicology test for cocaine or amphetamines at screening.

2. For participants of child bearing potential: breastfeeding, or positive urine pregnancy test prior to immunization or prior to CHMI.

3. Any history of malaria or previous participation in any malaria (vaccine) study or CHMI.

4. Known hypersensitivity to or contra-indications for both atovaquone/proguanil or artemether/lumefantrine. QT prolonging drugs are only considered an exclusion criterion when QT prolongation is observed at the ECG at screening.

5. A history of severe (allergic) reactions to mosquito bites. 6. Any history of infection with mycobacteria or BCG vaccination (only in stage B and C) 7. Any history of infection with yellow fever virus or yellow fever vaccination (only in stage B and C).

8. Participation in any other clinical study assessing an investigational medical product in the 30 days prior to the start of the study or during the study period.

9. Any condition or situation that could influence the independent consent of participant (e.g. being a direct colleague or family member of study personnel.

10. Any other condition or situation that would, in the opinion of the investigator, place the participant at an unacceptable risk of injury or render the participant unable to meet the requirements of the protocol or would compromise the integrity of the data.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Time to parasitemia | Moment of CHMI to antimalarial treatment (28 days post CHMI)
  The time to parasitemia (qPCR >100p/mL) (prepatent period) after CHMI in participants immunized with the GA2 parasite co-administered with an adjuvant compared to the unadjuvanted group and the infectivity controls.
Safety and tolerability: frequency and magnitude of adverse events in all study groups. | Moment of immunization to 35 days post CHMI
  The number of graded adverse events occurring in each group will be calculated as absolute numbers. Frequencies will be calculated by dividing the number of graded adverse events occurring in each group by the total number of volunteers in each group
Protective efficacy | Moment of CHMI to antimalarial treatment (28 days post CHMI)
  Proportion of participants immunized with the GA2 parasite co-administered with an adjuvant that do not develop parasitemia (qPCR >100p/mL) (sterile protection) after CHMI comparted the unadjuvanted group and the infectivity controls.

SECONDARY OUTCOMES:
Humoral immune responses of volunteers exposed to different intervention arms | Moment of immunization, pre-CHMI and up to 182 days post CHMI
  Difference in concentration of anti-CSP antibodies between intervention arms as assessed by ELISA.

OTHER OUTCOMES:
Cellular immune responses of volunteers exposed to different intervention arms | Moment of immunization, pre-CHMI and up to 182 days post CHMI
  Difference in percentage of CD4+ and CD8+ T-cells producing IFN-γ between intervention arms as assessed by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Meta Roestenberg, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roozen GVT, van Schuijlenburg R, Hensen ADO, Koopman JPR, Lamers OAC, Geurten FJA, Sijtsma JC, Baalbergen E, Janse JJ, Chevalley-Maurel S, Naar CM, Bezemer S, Kroeze H, van de Stadt HJF, de Visser B, Meij P, Tihaya MS, Colstrup E, Iliopoulou E, de Bes-Roeleveld HM, Wessels E, van der Stoep MYEC, Janse CJ, Murugan R, Franke-Fayard BMD, Roestenberg M. Single immunization with genetically attenuated Pf∆mei2 (GA2) parasites by mosquito bite in controlled human malaria infection: a placebo-controlled randomized trial. Nat Med. 2025 Jan;31(1):218-222. doi: 10.1038/s41591-024-03347-2. Epub 2025 Jan 3. PMID 39753962